CLINICAL TRIAL: NCT00477555
Title: Mosaic Ultra Porcine Bioprosthesis - Hemodynamic Study
Brief Title: Hemodynamic Assessment of Mosaic Ultra Stented Heart Valve in the Aortic Position
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: BRC-CS-14075
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Aortic Valve Replacement; Coronary Artery Bypass Grafting
Keywords: aortic valve; concomitant procedures; porcine bioprosthesis; stented valve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Aortic implantation of Mosaic Ultra porcine bioprosthesis — All patients get implanted with a Mosaic Ultra tissue valve to evaluate hemodynamic performance at 6 months post implant.

SUMMARY:
The special fixation methodology of the Mosaic Ultra stented procine bioprosthesis allows valves to maintain their natural leaflet structure and root geometry which prevents leaflet calcification and improves hemodynamic performance and a potential for increased durability. This study will document the hemodynamic performance, as assessed by echocardiographic recordings, at six months post implantation.

DETAILED DESCRIPTION:
1.0 STUDY PLAN 1.1. Study Objectives The objective of this clinical study is to evaluate the hemodynamic performance of the Mosaic Ultra™ stented porcine bioprosthesis in the aortic position.

1.2. Study Design This will be a prospective non randomized multi center clinical study designed to obtain hemodynamic data on the Mosaic Ultra™ stented porcine bioprosthesis. All participating centers follow a common clinical investigation plan.

1.3. Sample Size and Study Duration The basis for this study will be at least 60 MosaicÒ Ultra™ stented porcine bioprosthesis implants followed for six months.

2.0 PATIENT SELECTION 2.1. Patient Eligibility Criteria The patient population includes all patients who require aortic valve replacement for heart valve disease (acquired or congenital) and who are candidates for a bioprosthetic valve. Patients will be informed about the aspects of this study and will be asked to give their Informed Consent. The patient population must be geographically stable and able to attend one follow-up examination at the implanting center. Patients not willing or unable to fully participate in the follow-up will not be entered in the study.

2.2. Inclusion Criteria

* Patients who require aortic valve replacement with or without coronary artery bypass grafting or surgical treatment of Atrial Fibrillation.
* Patients who are able to provide informed consent.

3.3. Exclusion Criteria

* Concomitant procedures other than coronary artery bypass grafting or surgical treatment of Atrial Fibrillation.
* Patients indicated for receiving a mechanical prosthesis.
* Patients who will have a replacement of an existing valve prosthesis.
* Patients refusing or not able to provide informed consent.
* Patients requiring emergency surgery.

4.0 STUDY METHODS 4.1. Data Requirements For each patient enrolled in the study, information will be collected pre-operatively, operatively, and at 6 months post-operatively.

Patients entering the study are preoperatively evaluated for clinical information. Upon implant of the Mosaic bioprostheses the appropriate surgical data will be obtained. Follow-up data are required at discharge and six months post-operative. Endpoint for each patient in the study will be the six months follow-up.

The required variables are specified on each CRF. Samples of the CRF's are provided in Appendix C. Transthoracic echocardiography is required at pre-op and at six months.

All centers will be provided with a unique center ID. Enrolled patients will be identified on the CRF's by using the center ID with a sequential three digit number.

4.2. Case Report Form (CRF) Completion All appropriate sections of the case report forms must be filled out completely and accurately in black or blue ink. Before submission to Medtronic the investigator (or designated co-investigator) must review, sign and date the CRFs. The original is sent to Medtronic, and a copy remains at the center in the patient study file. All efforts should be made to submit CRFs to Medtronic within 6 weeks after the examination.

4.3. Study File A study file will be set up and maintained by the study center. This will be the repository for all records related to the study. All case report forms should be traceable to source documents. Source documents must be maintained in the patient medical records.

5.0 DATA ANALYSIS AND REPORTING 5.1. Data ownership All data collected in this study will be regarded as confidential and will be entered in a common database that is the property of Medtronic.

5.2. Data analysis Appropriate statistical analysis will be performed to compare the hemodynamic performance of various sizes. Hemodynamic data will be summarized by valve size. Descriptive statistics will be employed to report patient population characteristics, operative and post-operative data.

5.3. Data reporting Medtronic will complete and submit to the participating investigators a complete report using all collected data.

5.4. Publication policy It is the intent of both Medtronic and the study center that the investigator publish the results of this study. Medtronic may elect to use the data and outcomes of this study for the promotion of its products. Investigator will provide a copy of any abstract, presentation, and/or manuscript to Medtronic at least thirty (30) days prior to submission. Medtronic has the right to review the publications for confidential information, copyright materials and to edit for technical accuracy prior to submission.

6.0 STUDY MANAGEMENT 6.1. Study Sponsor and Contact Staff Medtronic Bakken Research Center B.V. is the sponsor of this study

Bèr Kleijnen, Sr. Clinical Research Specialist, will be the contact person for the overall study coordination:

Bèr Kleijnen Sr. Clinical Research Specialist Cardiac Surgery Clinical Operations Bakken Research Center B.V. Endepolsdomein 5 6229 GW Maastricht The Netherlands email:ber.kleijnen@medtronic.com

Your local Sales representative will be the contact person for the daily coordination and data collection:

6.2. Records Retention Records must be retained at each clinical site for a period of 2 years after the date the study is completed or terminated, and in accordance with local record retention requirement.

Medtronic will maintain clinical study records permanently. .

ELIGIBILITY:
Inclusion Criteria:

* Patients who require aortic valve replacement with or without coronary artery bypass grafting or surgical treatment of Atrial Fibrillation.
* Patients who are able to provide informed consent.

Exclusion Criteria:

* Concomitant procedures other than coronary artery bypass grafting or surgical treatment of Atrial Fibrillation.
* Patients indicated for receiving a mechanical prosthesis.
* Patients who will have a replacement of an existing valve prosthesis.
* Patients refusing or not able to provide informed consent.
* Patients requiring emergency surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are eligible for an aortic valve replacement can be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2006-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaak Minten, PhD, Study Director — Clinical Director Cardiac Surgery Medtronic
Locations (11):
- Medinische Universitat Innsbruck, Innsbruck, Austria
- Belgium (3):
  - ZNA Middelheim, Antwerp, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - Hopital St Luc, Bouge
- Germany (3):
  - Klinik fur Thorax- Herz und Gefasschirurgie, Dortmund
  - Klinikum der Johann-Wolfgang-Goethe Universitat, Frankfurt Am Mein
  - Albertinen Krankenhaus, Hamburg
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadasit Medical Research Services, Jerusalem
- U.O. Cardiochirurgia del p.p. Civico, Palermo, Italy